CLINICAL TRIAL: NCT02953808
Title: A Single Centre, Double-blind, Randomised, Placebo-controlled, and Single Dose-ascending Study to Investigate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics, of Single Intravenous Doses of GSK2315698 in Healthy Japanese Subjects
Brief Title: Phase 1 Study of GSK2315698 in Healthy Japanese Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 205911
Record Dates: First submitted 2016-11-01; First posted 2016-11-03 (Estimated); Last update posted 2017-01-19 (Estimated); Status verified 2017-01

CONDITIONS: Amyloidosis
Keywords: GSK2315698; Dose-ascending; Systemic amyloidosis
MeSH Terms: conditions — Amyloidosis; Immunoglobulin Light-chain Amyloidosis | interventions — miridesap

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (5):
- Cohort 1 Group A (Experimental): In dosing sessions 1, 2, and 3, subjects will receive GSK2315698 10 mg/hr, GSK2315698 20 mg/hr, and Placebo, respectively, as intravenous infusion over 1 hour.
  Interventions: Drug: Placebo; Drug: GSK2315698
- Cohort 1 Group B (Experimental): In dosing sessions 1, 2, and 3, subjects will receive GSK2315698 10 mg/hr, Placebo, and GSK2315698 40 mg/hr, respectively, as intravenous infusion over 1 hour.
  Interventions: Drug: Placebo; Drug: GSK2315698
- Cohort 1 Group C (Experimental): In dosing sessions 1, 2, and 3, subjects will receive Placebo, GSK2315698 20 mg/hr, and GSK2315698 40 mg/hr, respectively, as intravenous infusion over 1 hour.
  Interventions: Drug: Placebo; Drug: GSK2315698
- Cohort 2 Group D (Experimental): In a single dosing session, subjects will receive GSK2315698 20 mg/hr as intravenous infusion over 15 hours.
  Interventions: Drug: GSK2315698
- Cohort 2 Group E (Placebo Comparator): In a single dosing session, subjects will receive Placebo as an intravenous infusion over 15 hours.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Placebo — 0.9% weight by volume (w/v) saline solution for intravenous infusion over 1 hour (in Cohort 1) or over 15 hours (in Cohort 2).
  Arms: Cohort 1 Group A; Cohort 1 Group B; Cohort 1 Group C; Cohort 2 Group E
Drug: GSK2315698 — 200 mg/mL stock solution for intravenous infusion over 1 hour (in Cohort 1) or over 15 hours (in Cohort 2). The stock solution will be diluted to obtain dosage levels of 10 mg/hr, 20 mg/hr, or 40 mg/hr.
  Arms: Cohort 1 Group A; Cohort 1 Group B; Cohort 1 Group C; Cohort 2 Group D

SUMMARY:
This is the first study in which GSK2315698 will be administered in Japanese population. The primary objective of the study is to investigate safety and tolerability, pharmacokinetics, and pharmacodynamics after single intravenous infusion in healthy subjects. This will be a single center, double-blind, randomized, placebo-controlled, dose-ascending study.

Subjects in Cohort 1 will attend 3 dosing sessions, and will be randomized to one of the 3 groups. Each group will receive GSK2315698 and Placebo in a defined sequence. The dose levels of GSK2315698 are set to 10 milligrams (mg) per hour (hr), 20 mg/hr, and 40 mg/hr, to be administered over 1 hour. Dosing sessions 1 and 2, and dosing sessions 2 and 3, will be separated by a washout period of at least 8 and 10 days, respectively.

Subjects in Cohort 2 will attend a single dosing session, and will be randomized to receive either GSK2315698 20 mg/hr or Placebo, over a period of 15 hours.

A sufficient number of subjects will be randomized such that 18 subjects (9 in each cohort) complete the study. The duration of participation for any subject in this study will be approximately 59 days.

ELIGIBILITY:
Inclusion Criteria:

* Participant must be 20 to 64 years of age inclusive, at the time of signing the informed consent
* Participants who are overtly healthy as determined by medical evaluation including medical history, physical examination, laboratory tests, and cardiac monitoring. A subject with a clinical abnormality or laboratory parameter(s) which is/are not specifically listed in the inclusion or exclusion criteria, outside the reference range for the population being studied may be included only if the investigator in consultation with the Medical Monitor if required agree that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures
* Peripheral veins suitable for venous blood sampling and cannulation
* Body weight >=50 kilograms (kg) and body mass index (BMI) within the range 18.5-24.9 kg per meter (m) squared (inclusive)
* Male: A Japanese male participant must agree to use contraception during the treatment period and until follow up visit
* Capable of giving signed informed consent

Exclusion Criteria:

* History or presence of cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, hematological, or neurological disorders capable of significantly altering the absorption, metabolism, or elimination of drugs; constituting a risk when taking the study treatment; or interfering with the interpretation of data
* Clinically abnormal hypotonia or hyperpiesia as determined by the investigator
* Previous surgical procedures on the upper digestive tract including cholecystectomy (gallbladder removal), and/or cholelithotomy (gallstone removal)
* Alanine Aminotransferase (ALT) >1.5 multiplied by upper limit of normal (ULN)
* Bilirubin >1.5 times ULN (isolated bilirubin >1.5 times ULN is acceptable if bilirubin is fractionated and direct bilirubin <35%)
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones)
* QTcF >450 millisecond (msec) QTcF is either machine-read or manually over-read. The specific formula that will be used to determine eligibility and discontinuation for an individual subject should be determined prior to initiation of the study. In other words, several different formulae cannot be used to calculate the corrected QT interval (QTc) for an individual subject and then the lowest QTc value used to include or discontinue the subject from the trial. For purposes of data analysis, QTcF, another QT correction formula, or a composite of available values of QTc will be used
* Past or intended use of over-the-counter or prescription medication including herbal medications within 14 days prior to dosing. Specific study-defined medications may be allowed
* History of donation of blood or blood products >=400 mL within 3 months or >=200 mL within 1 month prior to screening
* Exposure to more than 4 new chemical entities within 12 months prior to the first dosing day
* Current enrollment or past participation within the last 3 months, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer) before signing of consent in this or any other clinical study involving an investigational study treatment or any other type of medical research
* The subject is positive for Serological test for syphilis (Rapid plasma reagin test [RPR] and Treponema pallidum Latex Agglutination [TPLA]), Human immunodeficiency virus (HIV) antigen/antibody, Hepatitis B surface antigen (HbsAg), Hepatitis C virus (HCV) antibody, or Human T-cell lymphotropic virus type 1 (HTLV-1) antibody at screening
* Positive pre-study drug screen
* Regular use of known drugs of abuse
* Regular alcohol consumption within 6 months prior to the study defined as an average weekly intake of >14 units for males. One unit is equivalent to 350 mL of beer, 150 mL of wine or 45 mL of 80 proof distilled spirits
* Smoking or history or regular use of tobacco- or nicotine-containing products within 6 months prior to screening; Sensitivity to any of the study treatments, or components thereof, or drug or other allergy that, in the opinion of the investigator or Medical Monitor, contraindicates participation in the study

Ages: 20 Years to 64 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2016-11; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Number of subjects with adverse events (AE) and serious adverse events (SAE) | Over a maximum period of approximately 29 days
Number of subjects with abnormalities in clinical laboratory parameters | Over a maximum period of approximately 59 days
  Abnormalities will be assessed in laboratory parameters of hematology, clinical chemistry, and routine urinalysis.
Number of subjects with abnormalities in vital sign parameters | Over a maximum period of approximately 59 days
  Abnormalities will be assessed in the vital signs of respiratory rate, pulse rate, blood pressure, and body temperature. Vital signs will be measured in a supine position after 5 minutes of rest.
Number of subjects with electrocardiogram (ECG) abnormalities | Over a maximum period of approximately 59 days
  Single 12-lead ECG will be obtained using an ECG machine that automatically calculates the heart rate and measures PR, QRS, QT, and QT interval corrected for heart rate by Fridericia's formula (QTcF) intervals.
Plasma concentration of GSK2315698 | Pre-dose and 0.25, 1, 2, 4, 6, 8, 12, 24 hours post-dose in Cohort 1; Day 1 (pre-dose and 0.25, 1, 4, 12, 15, 18, 24 hours post-dose), and Days 5, 8, 14 in Cohort 2
  Whole blood samples of approximately 2 milliliters (mL) will be collected for measurement of plasma concentrations of GSK2315698.
Maximum observed plasma concentration (Cmax) of GSK2315698 | Pre-dose and 0.25, 1, 2, 4, 6, 8, 12, 24 hours post-dose in Cohort 1; Day 1 (pre-dose and 0.25, 1, 4, 12, 15, 18, 24 hours post-dose), and Days 5, 8, 14 in Cohort 2
  Cmax will be calculated if data permit.
Area under the concentration-time curve from pre-dose to 24 hours (AUC0-24) of GSK2315698 | Pre-dose and 0.25, 1, 2, 4, 6, 8, 12, 24 hours post-dose in Cohort 1; Day 1 (pre-dose and 0.25, 1, 4, 12, 15, 18, 24 hours post-dose), and Days 5, 8, 14 in Cohort 2
  AUC0-24 will be calculated if data permit.
Time to maximum observed plasma drug concentration (Tmax) of GSK2315698 | Pre-dose and 0.25, 1, 2, 4, 6, 8, 12, 24 hours post-dose in Cohort 1; Day 1 (pre-dose and 0.25, 1, 4, 12, 15, 18, 24 hours post-dose), and Days 5, 8, 14 in Cohort 2
  Tmax will be calculated if data permit.
Cohort 2: Plasma concentration of GSK2315698 at 15 hours (C15hr) | Pre-dose and 0.25, 1, 4, 12, and 15 hours post-dose in Cohort 2
  C15hr will be calculated if data permit.
Change from Baseline in blood concentration of serum amyloid P component (SAP) | Day 1 (pre-dose and 0.25, 1, 2, 4, 6, 8, 12, 24 hours post-dose), Day 5, and Day 8 in Cohort 1; Day 1 (pre-dose and 0.25, 1, 4, 12, 15, 18, 24 hours post-dose), and Days 5, 8, 14 in Cohort 2
  Venous blood samples of approximately 2 mL will be collected for measurement of SAP.
Minimum blood concentration (Cmin) of SAP | Day 1 (pre-dose and 0.25, 1, 2, 4, 6, 8, 12, 24 hours post-dose), Day 5, and Day 8 in Cohort 1; Day 1 (pre-dose and 0.25, 1, 4, 12, 15, 18, 24 hours post-dose), and Days 5, 8, 14 in Cohort 2
  Cmin will be calculated if data permit.
Time to minimum observed concentration (Tmin) of SAP | Day 1 (pre-dose and 0.25, 1, 2, 4, 6, 8, 12, 24 hours post-dose), Day 5, and Day 8 in Cohort 1; Day 1 (pre-dose and 0.25, 1, 4, 12, 15, 18, 24 hours post-dose), and Days 5, 8, 14 in Cohort 2
  Tmin will be calculated if data permit.
Cohort 2: Concentration of SAP at 15 hours (C15hr) | Pre-dose and 0.25, 1, 4, 12, and 15 hours post-dose in Cohort 2
  C15hr will be calculated if data permit.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Tokyo, Japan